CLINICAL TRIAL: NCT05314985
Title: Effect of Preoperative Training and Education on Pre- and Postoperative Functional Performance in Patients Awaiting TKA; A Randomized Controlled Trial - a Pilot Study
Brief Title: Prehab Intervention in Patients Awaiting Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BASEC-Nr. 2020-03060
Record Dates: First submitted 2021-07-20; First posted 2022-04-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Preoperative Exercise; Physical Therapy Modalities; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehab Group / Intervention Group (Experimental): 4 to 8 weeks of preoperative physical therapy training and education intervention before total knee replacement surgery.
  Interventions: Other: Prehab intervention
- Control Group (No Intervention): Usual care / no treatment before total knee replacement surgery.

INTERVENTIONS:
Other: Prehab intervention — Individual training program containing strengthening, sensori-motor, joint mobilisation and endurance exercises as well as educational inputs concerning perioperative procedure and instructions on e.g. how to walk with crutches.
  Arms: Prehab Group / Intervention Group

SUMMARY:
The objectives of this study are to investigate the feasibility primarily and furthermore the effects of a four to eight-weeks program of a combined clinic- and home-based preoperative physical therapy (exercise training and education) versus usual care in patients awaiting unilateral primary TKA up to 3 months after surgery.

DETAILED DESCRIPTION:
The patients randomized into the intervention group are going to pass through a three-week therapy program. This program is based on MD's prescription and provides 9 sessions of physical therapy per prescription. All patients carry out their therapy at University Center for Prevention and Sports Medicine (UCePS) Balgrist. Before the evaluation phase starts, each patient is introduced by a member of the research team and gets a written information sheet about the goal of the study and the following procedure. The patients have to signature an informed consent to their participation in our investigation. Both groups are to be tested four times: The first assessment is appointed at a minimum of four weeks before surgery. Their baseline characteristics are noted, knee ROM, SCT, TUG, 5STS, 2MWT, handgrip strength and pain score are assessed and they need to fill in the KOOS, the Short Form 12 (SF-12) and the Tegner Activity Scale. After the first assessment, the Intervention Group (IG) is allowed to start the physical therapy exercise and education intervention. Each Physical Therapist treating a participant was previously introduced to the study protocol and the intended intervention. They conduct a total of 9 sessions over a 4 to 8-weeks period before surgery with one to two appointments per week. The Control Group (CG) is asked to keep its activity level as it is before the baseline measure. It is not desired, that anyone in this group starts a new type of therapy or training in preoperative stage. Patients in both groups keep their diary about changes concerning pain, medicament intake, training and therapies during the full length of intervention and follow-up phase.

One monitoring visit at the investigator's site prior to the start, one visit within one year after inclusion of the first participant and approximately once visit per annum during the course of the study will be organised by the Sponsor. Furthermore, there will be a monitoring visit at the study end. During the monitoring, all documents including source data/documents will be accessible for the monitor and all questions will be answered. Data will be entered in REDCap and retrieved from the clinic's information system.

If a subject is withdrawn, all previous collected data will be used for the final evaluation. All collected data will be used. An intention to treat analysis will be performed.

Data Handling and Record Keeping / Archiving:

* Case Report Forms (CRF): For each enrolled study participant, a printed CRF is maintained. Appropriate coded identification is used: Initials followed by birth year. CRF data is entered into an electronic database for analysis (double data entry).
* Specification of Source Documents: Source data is available at the site to document the existence of the study participants. Source includes the original documents relating to the study, as well as medical history of the participant. Source documents in this study are CRF, hardcopy of printed hearing thresholds (audiograms), informed consent forms and patient list. All hardcopies are collected in a file folder and stored in a lockable cabinet in the office of the PI.
* Record Keeping / Archiving: All study data is archived for a minimum of 10 years after study termination or premature termination of the clinical trial. All hardcopies are collected in a file folder and stored in a lockable cabinet in the office of the PI.

Data management:

* Data Management System: Data is entered in REDCap® electronic data capture system, provided by the University Hospital Balgrist.
* Data Security, Access and Back-up: Data is saved on the personal account. Backup system is in place and hosted by the IT department of the University Hospital Balgrist.
* Analysis and Archiving: Data is entered into an electronic database for analysis (SPSS).
* Electronic and Central Data Validation: All data collected for this research project will be registered in encrypted form in an automatic secure online processing (REDCap® electronic data capture system). Data entry is performed exclusively by authorized persons involved in the research project. Data processing and storage also takes place in REDCap®. Only encrypted data will be used for data analysis and statistical evaluation.

Reporting of Serious Adverse Events (SAE):

Clinical investigators and ultimately the Principal Investigator (PI) have the primary responsibility for SAE identification, documentation, grading, and assignment of attribution to the intervention under study. Clinical study participants will be routinely questioned about Adverse Events (AE) at study visits. The well-being of the participants will be ascertained by neutral questioning ("How are you?"). Observed or volunteered SAE, regardless of treatment group or suspected causal relationship to the study treatment(s) will be recorded in the patient file and subsequently in the electronic CRF (eCRF) if a relationship to the study intervention cannot be excluded. All SAEs in which a relation to the study intervention cannot be excluded, will be fully documented in the appropriate eCRF. For each such SAE, the investigator will provide the onset, duration, intensity, treatment required, outcome and action taken with the investigational device or study related procedure.The investigator shall report these events: a.) to the sponsor within 24 hours after they become known; and b.) to the responsible ethics committee via Business Administration System for Ethic Committees (BASEC) within 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female participants (≥18 years)
* Patients receiving a unilateral TKA
* Signed informed consent after being informed

Exclusion Criteria:

* BMI >35
* Patella alta (Caton Deschamps Index >1.2)
* Muscle weakness due to neurological diagnosis
* Known or suspected non-compliance
* Known depression or other psychiatric disorders
* Acute pain exacerbations or inflammation
* Patellar instability
* Contradictions on ethical grounds
* Non-German speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Preoperative functional performance compared to baseline | 2-10 days before sugery
  To compare functional performance immediately pre-surgery after preoperative physical therapy in patients awaiting a TKA to baseline.
  Assessment: Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.

SECONDARY OUTCOMES:
Preoperative functional performance compared to usual care | 2-10 days before sugery
  To compare functional performance immediately pre-surgery after preoperative physical therapy to patients with usual care.
  Assessment: Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.
Preoperative stair climbing before TKA compared to baseline | 2-10 days before sugery
  To compare stair climbing after preoperative physical therapy immediately pre-surgery to baseline in patients awaiting a TKA.
  Assessment is an indicator for stair climbing:
  - Stair Climbing Test (SCT)
Preoperative stair climbing before TKA compared to usual care | 2-10 days before sugery
  To compare stair climbing after preoperative physical therapy immediately before TKA to usual care.
  Assessment is an indicator for stair climbing:
  - Stair Climbing Test (SCT)
Preoperative walking performance before TKA compared to baseline | 2-10 days before sugery
  To compare walking performance after preoperative physical therapy immediately pre-surgery to baseline in patients awaiting a TKA.
  Assessment are indicators for walking performance:
  * 2-minute walking test (2MWT)
  * Timed-Up and Go (TUG)
Preoperative walking performance before TKA compared to usual care | 2-10 days before sugery
  To compare walking performance after preoperative physical therapy immediately pre-surgery to usual care in patients awaiting a TKA.
  Assessment are indicators for walking performance:
  * 2-minute walking test (2MWT)
  * Timed-Up and Go (TUG)
Preoperative strength before TKA compared to baseline | 2-10 days before sugery
  To compare strength after preoperative physical therapy immediately pre-surgery to baseline in patients awaiting a TKA.
  Assessments are indicators for strength:
  * 5-times Sit To Stand (5STS): indicator for knee strength
  * Handgrip Strength (HGS): indicator for strength of lower extremities
Preoperative strength before TKA compared to usual care | 2-10 days before sugery
  To compare strength after preoperative physical therapy immediately pre-surgery to usual care in patients awaiting a TKA.
  Assessments are indicators for strength:
  * 5-times Sit To Stand (5STS): indicator for knee strength
  * Handgrip Strength (HGS): indicator for strength of lower extremities
Preoperative activity level before TKA compared to baseline | 2-10 days before surgery
  To compare activity level before TKA to baseline.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Preoperative activity level beforeTKA compared to usual care | 2-10 days before surgery
  To compare activity level before TKA to patients with usual care.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Preoperative level of pain compared to baseline | 2-10 days before sugery
  To compare the level of pain after preoperative physical therapy immediately pre-surgery to baseline in patients awaiting a TKA.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Preoperative level of pain compared to usual care | 2-10 days before sugery
  To compare the level of pain after preoperative physical therapy immediately pre-surgery to patients with usual care.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Preoperative quality of life compared to baseline | 2-10 days before sugery
  To compare the quality of life after preoperative physical therapy immediately pre-surgery to baseline in patients awaiting a TKA.
  Assessment:
  - Short Form 12 (SF-12): The minimum score = 0, the maximum score = 100, where a higher score indicates a better outcome.
Preoperative quality of life compared to usual care | 2-10 days before sugery
  To compare the quality of life after preoperative physical therapy immediately pre-surgery to patients with usual care.
  Assessment:
  - Short Form 12 (SF-12): The minimum score = 0, the maximum score = 100, where a higher score indicates a better outcome.
Preoperative knee joint mobility compared to baseline | 2-10 days before surgery
  To assess preoperative range of motion (ROM) compared to baseline.
  Active knee joint mobility is assessed with a long-legged goniometer in supine position, where the patient pulls his/her heel towards his/her buttocks and extends his/her knee as far as possible.
  Assessment: Degrees [°] Notation: Neutral-zero-method
Preoperative knee joint mobility compared to usual care | 2-10 days before surgery
  To assess preoperative range of motion (ROM) compared to patients awaiting TKA with usual care.
  Active knee joint mobility is assessed with a long-legged goniometer in supine position, where the patient pulls his/her heel towards his/her buttocks and extends his/her knee as far as possible.
  Assessment: Degrees [°] Notation: Neutral-zero-method
Postoperative functional performance 6 weeks after TKA compared to baseline | 6 weeks postoperative
  To compare functional performance 6 weeks after TKA compared to baseline.
  Assessment:
  Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.
Postoperative functional performance 6 weeks after TKA compared to usual care | 6 weeks postoperative
  To compare functional performance 6 weeks after TKA to patients with usual care.
  Assessment:
  Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.
Postoperative activity level 6 weeks after TKA compared to baseline | 6 weeks postoperative
  To compare activity level 6 weeks after TKA to baseline.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Postoperative activity level 6 weeks after TKA compared to usual care | 6 weeks postoperative
  To compare activity level 6 weeks after TKA to patients with usual care.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Postoperative level of pain 6 weeks after TKA compared to usual care | 6 weeks postoperative
  To compare the level of pain 6 weeks after TKA to patients with usual care.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Postoperative level of pain 6 weeks after TKA compared to baseline | 6 weeks postoperative
  To compare the level of pain 6 weeks after TKA to baseline.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Feasibility of prehabilitation program: Number of participants with adherence to the therapy sessions of at least 80% | 6 weeks postoperative
  To assess feasibility of preoperative physical therapy intervention in patients awaiting a TKA (defined as adherence to the therapy sessions of at least 80%).
Dischargeability: Length of Stay in hospital (LoS) | 6 weeks postoperative
  To compare readiness for discharge from the hospital after surgery after preoperative physical therapy in patients awaiting a TKA to patients treated with usual care.
Postoperative functional performance 3 months after TKA compared to baseline | 3 months postoperative
  To compare functional performance 3 months after TKA to baseline.
  Assessment:
  Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.
Postoperative functional performance 3 months after TKA compared to usual care | 3 months postoperative
  To compare functional performance 3 months after TKA to patients with usual care.
  Assessment:
  Knee Osteoarthritis Outcome Score (KOOS). The minium score = 0 , the maximum score = 100, where a higher score indicates a better outcome.
Postoperative stair climbing 3 months after TKA compared to baseline | 3 months after sugery
  To compare stair climbing 3 months after TKA to baseline.
  Assessment is an indicator for stair climbing:
  - Stair Climbing Test (SCT)
Postoperative stair climbing 3 months after TKA compared to usual care | 3 months after sugery
  To compare stair climbing 3 months after TKA to usual care.
  Assessment is an indicator for stair climbing:
  - Stair Climbing Test (SCT)
Postoperative walking performance 3 months after TKA compared to baseline | 3 months after surgery
  To compare walking performance 6 weeks after TKA to baseline.
  Assessment are indicators for walking performance:
  * 2-minute walking test (2MWT)
  * Timed-Up and Go (TUG)
Postoperative walking performance 3 months after TKA compared to usual care | 3 months after surgery
  To compare walking performance 6 weeks after TKA to usual care.
  Assessment are indicators for walking performance:
  * 2-minute walking test (2MWT)
  * Timed-Up and Go (TUG)
Postoperative strength 3 months after TKA compared to baseline | 3 months after sugery
  To compare strength 3 months after TKA to baseline.
  Assessments are indicators for strength:
  * 5-times Sit To Stand (5STS): indicator for knee strength
  * Handgrip Strength (HGS): indicator for strength of lower extremities
Postoperative strength 3 months after TKA compared to usual care | 3 months after sugery
  To compare strength 3 months after TKA to ususal care.
  Assessments are indicators for strength:
  * 5-times Sit To Stand (5STS): indicator for knee strength
  * Handgrip Strength (HGS): indicator for strength of lower extremities
Postoperative activity level 3 months after TKA compared to baseline | 3 months postoperative
  To compare activity level 3 months after TKA to baseline.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Postoperative activity level 3 months after TKA compared to usual care | 3 months postoperative
  To compare activity level 3 months after TKA to usual care.
  Assessments:
  - Tegner Activity Scale (TAS): The minimum score = 0, the maximum score = 10, where a higher score indicates a better outcome.
Postoperative level of pain 3 months after TKA compared to baseline | 3 months postoperative
  To compare the level of pain 3 months after TKA to baseline.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Postoperative level of pain 3 months after TKA compared to usual care | 3 months postoperative
  To compare the level of pain 3 months after TKA to patients with usual care.
  Assessment:
  - Numeric rating scale (NRS): The minimum score = 0, the maximum score = 10, where a lower score indicates a better outcome.
Postoperative quality of life 3 months after TKA compared to baseline | 3 months postoperative
  To compare the quality of life 3 months after TKA compared to baseline.
  Assessment:
  - Short Form 12 (SF-12): The minimum score = 0, the maximum score = 100, where a higher score indicates a better outcome.
Postoperative quality of life 3 months after TKA compared to usual care | 3 months postoperative
  To compare the quality of life 3 months after TKA to patients with usual care.
  Assessment:
  - Short Form 12 (SF-12): The minimum score = 0, the maximum score = 100, where a higher score indicates a better outcome.
Postoperative knee joint mobility 3 months after TKA compared to baseline | 3 months after surgery
  To assess postoperative range of motion (ROM) 3months after TKA compared to baseline.
  Active knee joint mobility is assessed with a long-legged goniometer in supine position, where the patient pulls his/her heel towards his/her buttocks and extends his/her knee as far as possible.
  Assessment: Degrees [°] Notation: Neutral-zero-method
Postoperative knee joint mobility 3 months after TKA compared to usual care | 3 months after surgery
  To assess postoperative range of motion (ROM) 3 months after TKA compared to baseline.
  Active knee joint mobility is assessed with a long-legged goniometer in supine position, where the patient pulls his/her heel towards his/her buttocks and extends his/her knee as far as possible.
  Assessment: Degrees [°] Notation: Neutral-zero-method
Postoperative Global Impression of Change compared to usual care | 3 months after surgery
  To assess postoperative Global Impression of Change 3 months after TKA compared to usual care.
  Assessment: Patient Global Impression of Change (PGIC)-Score: The minimum score = 0, the maximum score = 7, where a lower score indicates a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Scherr, Prof., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make Individual Participant Data (IPD) available.

REFERENCES:
- [Derived] Granicher P, Kocher M, de Bie R, Swanenburg J, Scherr J. Exploring feasibility of health-related quality of life assessments and pain diaries in patients undergoing prehabilitation before total knee arthroplasty: a pilot study. BMC Musculoskelet Disord. 2025 Oct 23;26(1):988. doi: 10.1186/s12891-025-09184-9. PMID 41131492
- See also: Information on the prehabilitation program at University Hospital Balgrist. — https://www.balgrist.ch/angebot/zentren/zentrum-fuer-sportmedizin/praehabilitation/